CLINICAL TRIAL: NCT04273841
Title: Exploring the Impact of Sleep Deprivation and Caffeine on Operationally Relevant Complex Cognitive Processes in Medical Professionals
Brief Title: Impact of Sleep Deprivation and Caffeine in Medical Professionals
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Currently this study is unfunded, but WRAIR Principal Investigator (PI) and USUHS Site PI, will continue to search for restoral or Unfunded Requirement (UFR) funds that can resurrect this protocol and allow the opportunity to collect data.
Sponsor: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: WRAIR #2311
Record Dates: First submitted 2019-09-05; First posted 2020-02-18 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Sleep Deprivation; Performance
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Caffeine Group (Active Comparator): This group will receive caffeine gum.
  Interventions: Dietary Supplement: Military Energy Gum
- Placebo (Placebo Comparator): This group will receive gum without caffeine.
  Interventions: Dietary Supplement: Placebo Gum

INTERVENTIONS:
Dietary Supplement: Military Energy Gum — Caffeine (1, 3, 7-trimethylxanthine) is a central nervous system stimulant that is found naturally in some foods and beverages such as coffee and tea. For this study, caffeine will be administered in the form of gum pellets (Military Energy chewing gum). Each pellet contains 100 mg of caffeine.
  Arms: Caffeine Group
Dietary Supplement: Placebo Gum — Pellet form placebo gum
  Arms: Placebo

SUMMARY:
While the negative impact of sleep deprivation on cognitive processing and the partial reversal of this phenomenon by caffeine are well known, the types of cognitive processing previously studied have been limited to simple, straight-forward laboratory tasks. It is unclear how sleep deprivation and caffeine affect performance on operationally relevant complex cognitive tasks, like those encountered by working professionals such as doctors. This study aims to uncover how sleep deprivation and caffeine impact two types of clinical reasoning processes encountered by physicians on a daily basis. Previous work from members of our team investigated diagnostic reasoning in medical professionals and discovered that brain activation in executive processing areas was modulated by self-reported sleepiness and burnout and level of expertise (Durning, Costanzo, et al., 2013; Durning et al., 2014, 2015). The current study aims to expand upon those findings by also investigating a potentially more complex type of clinical reasoning, i.e. therapeutic reasoning, and directly manipulating sleep and caffeine use in a controlled sleep laboratory. Medical students, residents, and board-certified physicians will undergo thirty-seven hours of sleep deprivation and ten hours of sleep recovery in the sleep laboratory. During two FMRI scan sessions we will present high-quality validated multiple-choice questions on common patient situations in internal medicine to participants to explore brain activity during therapeutic reasoning compared with diagnostic reasoning. One FMRI scan will occur following a night of sleep deprivation, and another scan will occur following a night of recovery sleep. Additionally, half of the participants will receive caffeine gum during the sleep deprivation period, while the other half will receive placebo gum. This design will allow us to study the effect of sleep deprivation and caffeine on the neural correlates of diagnostic and therapeutic reasoning and performance in general.

ELIGIBILITY:
Inclusion Criteria:

1. Novice group --National Capital Area Interns and Medical Students (3rd and 4th year only)
2. Intermediate group - National Capital Area PGY-2 and 3 residents in internal medicine
3. Expert group-Board certified internists from National Capital Area

Exclusion Criteria:

Related to Sleep Research Center. The following exclusion criteria apply to all volunteers:

* Self-reported habitual nightly sleep amounts outside the target range of 6-9 hours (i.e., less than 6 hours per night or more than 9 hours per night, on average) (Post-consent Checklist)
* Self-reported nighttime lights-out times earlier than 2100 hours on average during weeknights (Sunday through Thursday) (Post-consent Checklist)
* Self-reported morning wake-up times later than 0900 on average during weekdays (Monday through Friday) (Post-consent Checklist)
* Self-reported habitual napping (> 4 time a week in conjunction with normal sleep habits) (Post-consent Checklist)
* Self-reported caffeine use in excess of 400 mg (e.g., approximately 8 caffeinated sodas or 4 12-oz cups of coffee) per day on average (Post-consent Checklist; document provides exclusionary limits for various caffeinated products).
* Score of lower than 31 or higher than 69 on the Morningness-Eveningness Questionnaire (MEQ form)
* Score of 14 or above on the Beck Inventory Form (BDI form)
* Score of 41 or above on the Spielberger Trait Anxiety Inventory
* History of cardiovascular disease (to include but not limited to arrhythmias, valvular heart disease, congestive heart failure, history of sudden cardiac death or myocardial infarction) (Medical History and Examination Form)
* History of neurologic disorder (to include, but not limited to epilepsy or another seizure disorder, amnesia for any reason, hydrocephalus, MS, narcolepsy or other sleep disorders) (Medical History and Examination form; sleep items on Post-Consent Checklist)
* Underlying pulmonary disease requiring daily inhaler use (Medical History and Examination form)
* Kidney disease or kidney abnormalities (Medical History and Examination form, laboratory results)
* Liver disease or liver abnormalities (Medical History and Examination form, laboratory results)
* Self-reported history of psychiatric disorder requiring hospitalization or psychiatric product for any length of time (Medical History and Examination form)
* Self-reported or suspected regular nicotine use or addiction, defined as more than 1 cigarette or equivalent per week, within the last 1 year (Medical History and Examination form)
* Self-reported or suspected heavy alcohol use; minimum limit to define heavy alcohol use is 14 drinks per week or as determined by the examining study licensed physician (Medical History and Examination form)
* Self-reported or suspected use of products or drugs that cannot be safely discontinued during in-laboratory phases, to be determined on a case-by-case basis by the examining study licensed physician (Medical History and Examination form)
* Self-reported or suspected current use of other illicit drugs, to include but not limited to benzodiazepines, amphetamines, cocaine, marijuana (Medical History and Examination form)
* Positive urine pregnancy result
* Female volunteers who are breastfeeding, lactating, or actively trying to conceive
* Resting blood pressure above 140/90 or resting pulse > 110 (Medical History and Examination form). Note that if a repeat measurement is within range then the volunteer will not be excluded.
* BMI ≥ 30 (Obese Class I or greater) (Medical History and Examination form)
* Clinically significant values (as determined by the reviewing study licensed physician) for any hematology or chemistry parameter. Reviewing physician may opt to repeat any clinically significant tests and include volunteers whose repeat test values are not clinically significant.
* Positive urine nicotine/cotinine result during screening visit (NicCheck™ I test strip results)
* Positive urine drug result during screening visit
* Any use of prescription or over-the-counter sleep aids during the 6 month period prior to screening indicative of a potential sleep disorder as determined by the examining study medical investigator [e.g., use of a sleep aid for several nights following time zone travel, or the occasional use of a sleep inducing medication (e.g. 1-2 times per month), would not necessarily constitute evidence of a sleep disorder and result in disqualification].
* Not fitting into one of four categories: 1) 3rd of 4th year medical student AND native English speaker, 2) medical intern, 3) PGY-2 or PGY-3 resident in internal medicine, 4) board-certified internist (Post-consent checklist)
* Inability to read and sign the consent and HIPAA authorization form
* Active duty military or federal personnel: not off duty and not on approved annual leave for the enrollment visit as well as the in-laboratory phase of the study

Related to FMRI task.

The following exclusion criteria apply to all subjects (MR Safety Screening form):

* The presence of incompatible shrapnel or implanted devices
* A history of prior inability to complete an MRI scan due to anxiety or claustrophobia (participants will not be able to take benzodiazepines or other sedatives prior to the scan to treat anxiety, as these would adversely impact thought processes).
* Being treated with calcium channel blocker medicines (because of the potential impact of such medicines on cerebral blood flow patterns).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-07-09 (Actual)

PRIMARY OUTCOMES:
Psychomotor Vigilance Task | 5 days
  Computer Based response time measurement
Clinical Reasoning Questions | 5 days
  Answer clinical board questions

SECONDARY OUTCOMES:
Actigraphy | 5 days
  Wrist movement and activity monitoring
Polysomnography | 5 days
  Measurement of brain activity
Structural Brain Scan-functional MRI | 5 days
  Measurement of structural brain topography to localize areas of functional activation using a functional MRI scan

CONTACTS AND LOCATIONS:
Locations (1):
- WRAIR Sleep Research Center, Silver Spring, Maryland, United States

IPD SHARING:
Plan to Share IPD: No